CLINICAL TRIAL: NCT05910489
Title: New Tools for the Detection of Micro and NanoPLastics (MNPLs) in Greenhouse Workers as a Population Highly Exposed to Plastics: Effect on Different Biomarkers of Genotoxic Effect
Brief Title: Micro and Nanoplastics in Greenhouse Workers: Biomarkers of Exposure and Effect
Status: Not yet recruiting | Type: Observational
Sponsor: Ricard Marcos (Other)
Collaborators: Instituto Murciano de Investigación Biosanitaria Virgen de la Arrixaca (Other); Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Sponsor-Investigator, Ricard Marcos, Professor, Universitat Autonoma de Barcelona
Organization: Universitat Autonoma de Barcelona (Other)
Other Study IDs: 2-1
Record Dates: First submitted 2021-11-30; First posted 2023-06-18 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Microplastics; Nanoplastics; Genotoxic Damage; Inflammation
Keywords: MNPLs; greenhouse workers
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Peripheral blood, urine, feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Biomonitoring studies to detect MNPLs in biological samples and study of health effects.
  Determination of MNPLs levels, genotoxic damage, and immunological effects
  Interventions: Other: Biomonitoring of MNPLs in biological samples of greenhouse workers and controls
- Greenhouse workers: Biomonitoring studies to detect MNPLs in biological samples and study of health effects.
  Determination of MNPLs levels, genotoxic damage, and immunological effects
  Interventions: Other: Biomonitoring of MNPLs in biological samples of greenhouse workers and controls

INTERVENTIONS:
Other: Biomonitoring of MNPLs in biological samples of greenhouse workers and controls — Detection of biomarkers of exposure and genotoxic effect in biological blood, urine, exhalated air condensate, and feces

SUMMARY:
MNPLs effects on human health are still preliminary. Workers exposed to plastic residues are exposed constantly to MNPLs. One of these jobs corresponds to greenhouse workers, that could be considered as a population highly exposed to plastics. The objective of the research is to be able to detect MNPLs on body fluids as well as their potential genotoxic and immunological damage.

DETAILED DESCRIPTION:
The exponential increase in the production/use of plastic translates into a parallel increase of environmental plastic waste that is continuously degraded into MNPLs. Information on the MNPLs' effects on human health is still preliminary and, furthermore, the limitations in current methodologies prevent accurate exposure/risk assessment.

This observational study will obtain body samples of greenhouse workers and from a control group. That would allow optimizing specific biomarkers of human MNPLs exposure and the characterization of biomarkers of early effect that allows an association among the exposure to MNPLs and effects on human health.

ELIGIBILITY:
Inclusion Criteria of workers exposed to plastic residues:

* Working in an operating greenhouse for a period of 1 month or more
* Age over 18 years old
* Absence of chronic pathology including neoplasia
* Absence of infectious disease at the date of sample collection and for a period of more than 2 weeks
* Spanish residence

Inclusion Criteria of controls :

* Age over 18 years old. Matched by age, gender, and lifestyle to the exposed group.
* Absence of chronic pathology including neoplasia
* Absence of infectious disease at the date of sample collection and for a period of more than 2 weeks
* Spanish residence

Exclusion Criteria of workers exposed to plastic residues:

* Participation in another clinical study
* Pregnancy
* Unsigned informed consent

Exclusion Criteria of controls:

* Participation in another clinical study
* Pregnancy
* Unsigned informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will study adult professionals working in greenhouses in the countryside of Cartagena and Almeria. At least 25 volunteer professionals willing to participate in the study will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Biomonitoring study to detect the presence of MNPLs in body fluids | Up to 1 year
  Blood, buccal cells, exhalate breath condensate, feaces and urine will be collected from donors to check for the presence of micro and nanoplastics and/or derivatives
Genotoxicity effects of exposure to MNPLs | Up to 1 year
  Blood and buccal cells will be collected from donors to check for the presence genotoxic permanent damage, assessed by the micronucleus assay
Genotoxicity effects of exposure to MNPLs | up to 1 year
  Blood will be collected from donors to check for the presence genotoxic non-permanent damage, assessed by the comet assay
Study of the effects of MNPLs on immune system | Up to 1 year
  Blood will be collected from donors to check if the presence of micro and nanoplastics have an effect on th function of the immune system (signalling and activation) in vivo and in high-risk individuals

SECONDARY OUTCOMES:
Surrogate biomarkers after MNPLs exposure | Up to 1 year
  If it is possible to correlate the presence of micro and nanoplastics with the presence of plastic derivatives in body fluids, as blood or urine, this will facilitate the detection of plastic, because tecniques to detect surrogate biomarkers as e.g. plasticizers or antioxidants are cheaper and most use than the tecnology to detect MNPLs. For that different analytical tecniques will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Pelegrín, Principal Investigator — Instituto Murciano de Investigación Biosanitaria (IMIB); Juan Bernardo Cabezuelo, Study Chair — Hospital Clínico Universitario Virgen de Arrixaca (Murcia); Laura Martínez, Study Chair — Hospital Clínico Universitario Virgen de Arrixaca (Murcia)